CLINICAL TRIAL: NCT06665204
Title: Evaluating the Effectiveness of Clinical Practice Guideline Adherence for Patellofemoral Pain (knEE-CAPP)
Brief Title: Evaluating the Effectiveness of Clinical Practice Guideline Adherence for Patellofemoral Pain
Acronym: knEE-CAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Gorczynski (U.S. Federal Agency)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); University of Pittsburgh (Other); Chapman University (Other); The Geneva Foundation (Other); Naval Hospital Camp Pendleton (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor-Investigator, Sara Gorczynski, Research Physical Therapist, United States Naval Medical Center, San Diego
Organization: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMCSD.2024.0040; CDMRP-OR230100 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Patellofemoral Pain
Keywords: Physical Therapy; Military; Service members; Rehabilitation; Clinical Practice Guidelines
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Upon completing the informed consent, eligible participants will complete baseline questionnaires, then be randomized to 1) a CPG-adherent (intervention) arm in which PFP care is provided by research physical therapists based on CPG recommendations, and 2) a UC (comparator) arm, in which management decisions are made by non-research physical therapists in alignment with their personal and organizational practice standards but with no specific directives from the research team.
Who Masked: Participant
Masking Description: Given the nature of the CPG-adherent and UC intervention arms, it is not possible to blind treating physical therapists to treatment assignments; however, study participants will be blinded to their group assignments. Research personnel will be trained to endorse clinical equipoise of the two intervention arms during the informed consent process to limit unintentional biases.
  Further, all baseline and follow-up assessments will be administered remotely and distributed by a research team member who was not present for the study intervention (i.e., physical therapy treatment), limiting the potential influence of unblinded assessors on the outcomes of the study. Research team members facilitating remote baseline and follow-up assessments will be instructed to not answer or provide any direct guidance regarding completion of patient-reported outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Practice Guideline-adherent Care (Experimental): Participants randomized to receive CPG-adherent care will first receive a comprehensive clinical examination following the PFP CPG Decision Tree guidelines. Their treatment plan of care will correspond to any and all impairment subcategories, as defined by the PFP CPG.
  Interventions: Other: Clinical Practice Guideline-adherent Care
- Usual Care (Active Comparator): All participants randomized to the UC group will receive routine physical therapy evaluations and treatments in the outpatient physical therapy clinics at each participating military treatment facility, at the discretion of the staff physical therapist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Clinical Practice Guideline-adherent Care — Clinical examination procedures will be used to identify all appropriate impairment subcategories (Overuse/Overload without Other Impairment, PFP with Movement Coordination Deficits, PFP with Muscle Performance Deficits, PFP with Mobility Impairments) and create a subcategory-specific or multimodal (for patients classified to >1 subcategory) plan of care. Research physical therapists will target all applicable impairment subcategories using the corresponding CPG-recommended interventions, all of which are recommended for use as part of standard-of-care physical therapy practice. The duration and length of care will not be prespecified or standardized across participants to allow flexibility pending participant's care needs and schedule (e.g., vacation, short-term TDY status); however, research PTs will be trained to target providing no more than 10-12 visits over no more than 6-8 weeks to promote generalizability of the CPG-adherent intervention.
  Other Names: CPG-adherent Care
  Arms: Clinical Practice Guideline-adherent Care
Other: Usual Care — Usual physical therapy care will be provided by a licensed outpatient staff physical therapist who is not associated with the research team. The outpatient physical therapists will not treat participants in the CPG-adherent group and will be free to treat their participants based on their current personal and organizational clinical practice standards. The research team will neither influence nor restrict the evaluations conducted or interventions provided.
  Other Names: Usual physical therapy care
  Arms: Usual Care

SUMMARY:
The overall goal of this multisite, randomized clinical trial is to evaluate the short- and long-term effectiveness of a Clinical Practice Guideline (CPG)-adherent physical therapy approach to patellofemoral pain (PFP) management among military Service members. The main questions it aims to answer are:

1. Can a CPG-adherent care approach to PFP management improve short- and long-term knee function, pain, and confidence with completing duty-related activities?
2. Can a CPG-adherent care approach to PFP management reduce utilization of healthcare resources and analgesic medication prescription at 12-month follow-up?
3. Are there patient- and care-specific factors that predict or mediate clinical benefit from physical therapy care for PFP?

Researchers will compare the CPG-adherent physical therapy intervention to usual physical therapy care in the Military Health System.

Participants will: 1) be randomized to receive CPG-adherent care or usual care for PFP management; 2) attend physical therapy corresponding to their group assignment; and 3) complete patient-reported outcome measures at baseline and 6-weeks and 3-, 6-, and 12-months post-randomization.

DETAILED DESCRIPTION:
Knee injuries are among the most common musculoskeletal injuries affecting military personnel, accounting for 22% of limited duty profiles and an average of 53 limited duty days per injury in 2017 alone. Patellofemoral pain (PFP) is the most prevalent knee injury affecting Service members but has historically been considered an innocuous and self-limiting condition despite its high rate of persistence. Physical therapy is often the first line-of-defense for PFP management. Published data support the notion that adherence to evidence-based Clinical Practice Guidelines (CPG) improves outcomes 1) for patients, via greater improvements in pain and disability; 2) for providers, by supporting clinical decision making and practice efficiency; and 3) for healthcare systems, by reducing length of treatment, resource utilization, and costs. In 2019, the American Physical Therapy Association (APTA) published its first CPG for PFP management to better enable physical therapists to make evidence-based treatment decisions; however, there is limited evidence regarding the effectiveness of a collective, standardized CPG-adherent approach in clinical care. To evaluate whether patients with PFP who receive CPG-adherent care demonstrate superior outcomes as compared to patients receiving the current usual care, we will compare: (1) CPG-adherent care (intervention arm), wherein physical therapy care is provided according to the CPG "Decision Tree" recommendations for PFP management, to (2) Usual Care (UC; comparator arm), wherein care decisions are made by non-research physical therapists in alignment with current organizational and clinical practice standards in the Military Health System (MHS). This multisite, single-blind randomized controlled trial will include 440 active-duty Service members with PFP across four major MHS physical therapy facilities (i.e., Naval Medical Center San Diego, Naval Hospital Camp Pendleton, Brooke Army Medical Center, and Womack Army Medical Center). The sample will include Service members from the Army, Navy, and Marines, as well as both conventional and special operations forces. The co-primary outcomes include changes in two CPG-recommended outcome measures [Anterior Knee Pain Scale (AKPS) and the Numeric Pain Rating Scale (NPRS)]. Outcomes will be assessed at baseline; 6-weeks post-randomization; and 3-, 6-, and 12-months post-randomization (primary endpoint: 3-months). Secondary outcomes will include between-group differences in confidence with completing duty-related tasks and 12-month analgesic medication prescription and PFP-specific medical resource utilization. An exploratory analysis will seek to determine the predictors and mediators of clinical benefit from physical therapy care for Service members with PFP. Baseline and follow-up assessments will be administered remotely to maximize participant reach and retention. The intervention of interest, CPG-adherent care, is designed to be clinically feasible, with high potential for clinician adoption, which may improve care quality and patient outcomes for Service members with PFP. Long-term, findings from this study have the potential to improve patient care for PFP and other musculoskeletal injury conditions across the MHS by demonstrating the feasibility and positive impact of CPG-adherent care, particularly in terms of improving clinical outcomes and resource utilization and reducing unwanted variability in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty Service member
* Aged ≥18 years
* Presence of unilateral or bilateral PFP based on the core criterion of peripatellar and/or retropatellar pain with reproduction of PFP by at least one activity that loads the patellofemoral joint during weight bearing on a flexed knee, such as prolonged sitting, kneeling, squatting, hopping, running, stair climbing, patellar palpation
* Available to participate in physical therapy treatment within 6 weeks of initial enrollment

Exclusion Criteria:

* Presence of tibiofemoral OA based on imaging evidence in the electronic health records in the past year or self-report
* History of patellar or intra-articular knee trauma (e.g., dislocation/fracture) or surgery
* History of neurodegenerative conditions that may affect movement patterns (e.g., Multiple Sclerosis)
* Meniscal or ligamentous pathologies within the past year based on imaging evidence of acute injury in the electronic health record or self-report
* Quadriceps or patellar tendon injuries within the past year based on imaging evidence of acute injury in the electronic health record or self-report
* Known pregnancy (pregnant females may be eligible for participation after end of pregnancy and medical clearance by a qualified and licensed healthcare provider)
* Receipt of physical therapy care for PFP within the three months prior to enrollment
* Known to be pending medical evaluation board, discharge from the military, scheduled deployment, or litigation for an injury at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2027-09-29 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Anterior Knee Pain Scale (AKPS) | 6-weeks, 3-months (primary endpoint), 6-months, and 12-months post-randomization
  The AKPS is a CPG-recommended, 13-item questionnaire assessing knee function in people with PFP, with items differentially weighted for a maximum score of 100 and higher scores indicating better function.
Numeric Pain Rating Scale (NPRS) | 6-weeks, 3-months (primary endpoint), 6-months, and 12-months post-randomization
  The 11-point NPRS is a CPG-recommended measure of pain intensity in which patients rate their pain ranging from 0 (no pain) to 10 (worst imaginable pain).24-26 Average pain intensity in the past week will be assessed as part of the 3-item PEG, which includes 1-item each regarding average pain intensity, pain interference with enjoyment of life, and impact of pain on general activity.

SECONDARY OUTCOMES:
Perceived Duty-related Confidence | 6-weeks, 3-months, 6-months, and 12-months post-randomization
  Perceived confidence with completing duty-related activities will be evaluated using four questions assessing confidence with and perceived ability to perform military-related tasks, two of which are pulled from the Military Orthopedics Tracking Injuries and Outcomes Network (MOTION) Readiness Rehab questionnaire.
12-month Healthcare Utilization | 12-months post-randomization
  We will use individual electronic health record reviews alongside readily available EHR data elements indexed within Military Health System databases to determine the type and frequency of services received related to knee care during the 12 months following randomization. All medical resource utilization data will be identified and categorized using Healthcare Common Procedure Coding System (HCPCS) Level 1 current procedural terminology (CPT) 4 and 2 codes, International Classification of Disease, 10th Revision (ICD-10) codes, Medical Expense and Performance Reporting System (MEPRS) codes, and/or Health Insurance Privacy Authorization Act (HIPAA) taxonomy numbers. The categories that will be compared include: 1) visits to specialist clinics (e.g., sports medicine, orthopedists, physiatrists, pain management) and other health care providers, 2) diagnostic tests (e.g., x-rays, magnetic resonance imaging), and 3) surgical procedures.
12-month Analgesic Prescription | 12-months post-randomization
  Medication prescription will be queried using the Pharmacy Data Transaction Service. All medications prescribed to each patient during the 12-month follow-up period (beginning with randomization) will be reviewed. For those identified as analgesics, details such as product name, therapeutic and generic classes, number of days' supply, fill date, and dosage will be extracted to characterize the total number of unique analgesic prescriptions, total days' supply, and days to last prescription during the surveillance period.

OTHER OUTCOMES:
Optimal Screening for Prediction of Referral and Outcome Yellow Flag Assessment Tool - 10-item (OSPRO-YF) | 6-weeks and 3-months post-randomization
  The Optimal Screening for Prediction of Referral and Outcome Yellow Flag (OSPRO-YF) Assessment Tool is a multidimensional psychological assessment tool that has been used to identify psychological phenotypes associated with pain-related health outcomes (e.g., functional disability, sleep disturbance, catastrophizing). The OSPRO-YF can accurately estimate patient scores on a variety of validated, full-length outcome measures assessing pain-related psychological function (e.g., Pain Catastrophizing Scale, Tampa Scale of Kinesiophobia, Pain Self-efficacy Questionnaire) and identify whether scores reflect a "yellow flag" (i.e., surpass prognostic thresholds for development of disability after musculoskeletal pain onset).
Global Rating of Change (GROC) | 6-weeks, 3-months, 6-months, and 12-months post-randomization
  Global Rating of Change (GROC) is a one-item, 15-point scale, that provides information about self-perceived improvement in a patient ranging from -7 (a very great deal worse) to +7 (a very great deal better) with 0 in the middle (about the same). Scores of +4 and +5 are indicative of moderate changes in status, while +6 and +7 are indicative of a large change in a person's status.
Patient-reported Outcomes Measurement Information System (PROMIS) Computer Adaptive Tests (CATs) | 6-weeks, 3-months, 6-months, and 12-months post-randomization
  The Physical Function and Pain Interference CATs will be included, which are intended for clinicians and researchers in various disciplines who are interested in measuring physical, mental, and social health among individuals with various chronic conditions. All PROMIS® scores are reported on a T-score metric, where T-score of 50 aligns with the general population mean (standard deviation: 10). Higher scores indicate more of the domain being assessed.
Pain Sensitivity Questionnaire | 6-weeks, 3-months, 6-months, and 12-months post-randomization
  The Pain Sensitivity Questionnaire (PSQ)49 is designed to assess sensitivity to pain by asking participants to rate the pain intensity they would imagine experiencing in everyday pain-inducing scenarios. It includes 17 items rated from 0-10, where a score of '10' indicates the most painful sensation. The total score is calculated by summing each item with the exceptions of 5, 9, and 13 (as these situations do not reflect painful situations). The PSQ is a validated outcome measure that is predictive of sensitivity to experimental pain thresholds for mechanical, heat, and cold pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Gorczynski, PT, DPT, Study Director — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The final trial dataset will be made available to the research community upon request to and review by the Leadership Team. Data sharing agreements will be established to document the conditions for research use, privacy and confidentiality standards at the recipient site, and prohibitions for manipulating data for the purposes of identifying individuals. The final trial dataset will include all coded participant data (i.e., data that is de-identified by use of a unique study identification variable, with removal or modification of all identifiers). Individual-level data will include all screening information, baseline measures, intervention information, and primary and secondary outcomes. All SAS datasets will be supplied via secure transfer with the study protocol and data documentation (procedures used to collect the data, details about codes, variable definitions, variable field location, and type of variable).
Supporting Information: Study Protocol, SAP
Time Frame: Datasets will be available no later than the acceptance for publication of the primary and secondary findings from the final data set or one year after database lock.